CLINICAL TRIAL: NCT03045016
Title: Preliminary Study About the Efficacy of an α1 Blocker (Prazosin) in Preventing the Occurrence of Post-traumatic Stress Disorder (PTSD) in Patients With Acute Stress
Brief Title: Efficacy of Prazosin in Preventing Post-traumatic Stress Disorder
Acronym: PRAZOSTRESS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL16_0628
Record Dates: First submitted 2017-02-02; First posted 2017-02-07 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Acute Stress Disorder
Keywords: Acute stress Disorder; Post Traumatic Stress Disorder; Prevention; trauma; prazosin
MeSH Terms: conditions — Stress Disorders, Traumatic, Acute; Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Prazosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prazosin, ALPRESS® LP 2,5 et 5 mg (Experimental): Patients included in this study will be adults with acute stress as a result of a direct experience traumatic event. They will be treated with Prazosin, ALPRESS® LP 2,5 et 5 mg during 28 days.
  Interventions: Drug: Prazosin, ALPRESS® LP 2,5 et 5 mg

INTERVENTIONS:
Drug: Prazosin, ALPRESS® LP 2,5 et 5 mg — Patients will take Prazosin during 28 days ; there are two periods of treatment (escalation of doses):
  * PERIOD 1 (Day 0 - Day 7): 1 tablet of ALPRESS LP 2.5 mg (Prazosin) at bedtime for 7 days
  * PERIOD 2 (Day 8 - Day 27): 1 morning tablet of ALPRESS LP 5 mg (Prazosin) at bedtime for 21 days.

SUMMARY:
After a traumatic event such as an accident or an assault, victims may experience intense stress symptoms that may evolve into "post-traumatic stress disorder" (PTSD). It is a frequent and serious pathology, which can be complicated by depression, addiction or suicide. Few means are available to prevent PTSD in people who have just undergone trauma. Prazosin is an antihypertensive drug that blocks α1 adrenaline receptors which could help to stop the vicious circle of stress and prevent the development of the disease. The objective of this study is to demonstrate the efficacy of prazosin to prevent PTSD in patients who visit an emergency department after trauma.

ELIGIBILITY:
Inclusion Criteria:

* Patient of age >18 years and <65 years
* Victim of direct experience trauma (accident or physical aggression)
* Presence of an ASD between D3 and D7 after the trauma according to DSM V criteria

Exclusion Criteria:

* Contra-indication to prazosin: orthostatic hypotension, right heart failure, other hypotensive therapy, 5-phosphodiesterase inhibitors (sildenafil) or diuretic, history of syncope or severe unexplained faintness, hypersensitivity known to quinazolines.
* Alcohol and / or drug use at the time of the trauma
* History of psychotic disorder
* Suicidal risk defined by a score ≥ 2 on the Suicidal Ideas Item of the Beck Depression Inventory (BDI)
* Protected or vulnerable Major
* Persistence of a life threatening injury at D3
* Sexual assault
* Only moderate head trauma can be included and therefore excluded patients with loss of consciousness greater than 30 minutes, Glasgow score less than 13, post-traumatic amnesia greater than 24 hours (Ruff et al., 2009) .
* Prescription of morphine or morphine derivative in progress
* Pregnancy or breastfeeding period
* Lack of effective contraception in a woman susceptible to childbearing
* Known hepatic dysfunction
* Narcolepsy (Gelineau's disease)
* Cardiac or vascular history including coronary artery disease
* Strict low-sodium diet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
PTSD diagnosis | 6 months
  The Presence of PTSD diagnosis will be assessed by the Clinician Administered PTSD Scale (CAPS)

SECONDARY OUTCOMES:
Acute stress symptoms | 14 days
  These symptoms are assessed by Diagnostic and Statistical Manual of Mental Disorders (DSM V) criteria
Prazosin side effects | 7 days
  This will be investigated using a self questionnaire about frequent side effects due to Prazosin, measurement of blood pressure, and orthostatic hypotension test
Prazosin side effects | 14 days
  This will be investigated using a self questionnaire about frequent side effects due to Prazosin, measurement of blood pressure, and orthostatic hypotension test
Prazosin side effects | 1 month
  This will be investigated using a self questionnaire about frequent side effects due to Prazosin, measurement of blood pressure, and orthostatic hypotension test
occurrence of complications of PTSD | 6 months
  Complications of PTSD are attempted suicide, suicidal ideation, addiction, depression and quality of life.
Compliance | 1 month
  Compliance will be evaluated by counting the tablets consumed and not consumed at the end of the treatment by Prazosin

CONTACTS AND LOCATIONS:
Locations (1):
- Groupement Hospitalier Edouard Herriot - Emergency Psychiatry Department, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Magnin C, Poulet E, Fanton L, Vignaud P, Brunelin J. A non-randomized pilot trial of the use of prazosin in the prevention of transition from acute stress disorder to post-traumatic stress disorder. Eur J Psychotraumatol. 2023;14(2):2251250. doi: 10.1080/20008066.2023.2251250. Epub 2023 Sep 6. PMID 38154074